CLINICAL TRIAL: NCT04662216
Title: Clinical and Microbiological Efficacy of Chloramine and Hyaluronic Acid Gels in Non-surgical Periodontitis Treatment: a Randomized Controlled Clinical Trial
Brief Title: Clinical and Microbiological Efficacy of Chloramine and Hyaluronic Acid Gels in Non-surgical Periodontitis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Egle Ramanauskaite, pHd student, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol1, Version2
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Periodontitis
Keywords: periodontitis; scaling and root planing; sodium hypochlorite
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: The treatment will consist of two treatment modalities: (1) Control group - full mouth scaling and root planing (SRP) (2) Test group - full mouth SRP + "Perisolv" +"Hyadent BG" gels.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Periodontal examination, microbiologic sampling and professional oral cleaning will be performed by the investigator, unaware of periodontal treatment. Periodontal treatment will be performed by the investigator, unaware of clinical examination. Microbiological analysis will be performed by a third investigator, masked from clinical measurements and periodontal treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Scaling and root planing
  Interventions: Procedure: Scaling and root planing + "Perisolv" +"Hyadent BG" gels
- test group (Experimental): scaling and root planing + "Perisolv" +"Hyadent BG" gels.
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — Scaling and root planing will be accomplished with ultrasonic and hand instruments (Gracey curettes).
  Arms: test group
Procedure: Scaling and root planing + "Perisolv" +"Hyadent BG" gels — Scaling and root planing will be accomplished with ultrasonic and hand instruments (Gracey curettes), "Perisolv" gel will adjectively be applied to all pockets with probing depth(PD) ≥ 5 mm, which will be inserted into periodontal pockets before and during SRP (2 times). The nozzle will be placed in the pocket mesially, lingually, distally and bucally. Afterwards, all teeth will be polished and all treated pockets will be filled with hyaluronic acid gel (Hyadent BG).
  Arms: control group

SUMMARY:
The aim of the study is to investigate clinical and microbiological effects of subgingival application of chloramine (Perisolv) and hyaluronic acid (Hyadent BG) gels as adjuncts to scaling and root planing in non-surgical periodontitis treatment.

DETAILED DESCRIPTION:
Objectives:

1. To evaluate if additional subgingival delivery of chloramine and hyaluronic acid gels would enhance clinical outcomes of scaling and root planing in periodontitis patients.
2. To assess if additional subgingival delivery of chloramine and hyaluronic acid gels would reduce total counts of periodontopathogenic bacteria compared to scaling and root planing alone.

The treatment will consist of two treatment modalities: (1) Control group - full mouth scaling and root planing (SRP) (2) Test group - full mouth SRP + "Perisolv"+ Hyadent BG gels.

The periodontal treatment will be performed in one session without time restrictions. Under local anesthesia, an experienced operator, will perform a full mouth subgingival scaling and root planing with an ultrasonic device and Gracey curettes. Afterwards, all teeth will be polished using a low-abrasive paste.

Teeth in the test group (all teeth with PD ≥ 5 mm) will adjunctively be treated with chloramine gel (Perisolv), which will be inserted into periodontal pockets before and during SRP (2 times). The nozzle will be placed in the pocket mesially, lingually, distally and bucally. Teeth will be polished and all treated pockets will be filled with hyaluronic acid gel.

Teeth in control group will receive SRP + polishing

ELIGIBILITY:
Inclusion Criteria:

* > 30 years old;
* Good general health according to medical history and clinical judgment;
* Exhibiting at least one pocket in each quadrant with pocket depth (PD) ≥ 5 mm;
* Radiographic evidence of bone loss ( > 2 mm from cemento-enamel junction (CEJ) );
* Untreated periodontal disease;
* Minimum 20 teeth (wisdom teeth excluded);
* No removable prosthesis.

Exclusion Criteria:

* Patients already included in other clinical trials;
* Periodontal treatment during the last 12 months;
* Antibiotic treatment 6 months prior to the start of the trial;
* Antibiotic prophylaxis required for dental treatment;
* Ongoing medication that may affect the clinical features of periodontitis;
* Pregnant/lactating.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Probing depth (PD) reduction | 6 months
  PD (probing depth): the distance (mm) between the gingival margin and the bottom of the sulcus/pocket

SECONDARY OUTCOMES:
Clinical attachment level (CAL) | 6 months
  CAL (clinical attachment level): will be calculated for each site as the sum of PD and the gingival recession/overgrowth.
Bleeding on probing (BOP) | 6 months
  BOP (bleeding on probing): presence (+) or absence (-) of bleeding within 15s after probing the pocket (%).
Plaque Index (PI) | 6 months
  PI (Plaque index): presence of dental plaque along the mucosal margin at 6 sites of the implant presence (+) or absence (-).
Reduction of total counts of periodontopathogenic bacteria | 6 months
  Subgingival plaque samples will be analyzed for Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia Treponema denticola and Prevotella intermedia

CONTACTS AND LOCATIONS:
Overall Officials: Vita Machiulskiene, Prof, Study Chair — LUHS
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Kauno, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramanauskaite E, Machiulskiene V, Shirakata Y, Dvyliene UM, Nedzelskiene I, Sculean A. Clinical evaluation of sodium hypochlorite/amino acids and cross-linked hyaluronic acid adjunctive to non-surgical periodontal treatment: a randomized controlled clinical trial. Clin Oral Investig. 2023 Nov;27(11):6645-6656. doi: 10.1007/s00784-023-05271-0. Epub 2023 Sep 23. PMID 37740107